CLINICAL TRIAL: NCT06606340
Title: A Long-term Observational Study Evaluating Sarepta Therapeutics, Inc.'s Exon-Skipping Therapies in Patients With Duchenne Muscular Dystrophy Under Conditions of Routine Clinical Practice
Brief Title: A Long-term Observational Study Evaluating Eteplirsen, Golodirsen, or Casimersen in Routine Clinical Practice
Acronym: EVOLVE
Status: Enrolling by invitation | Type: Observational
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 4658-403
Record Dates: First submitted 2024-08-08; First posted 2024-09-23 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; DMD; Post-marketing; Observational; Phase 4; Eteplirsen; Golodirsen; Casimersen
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen; golodirsen; casimersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Eteplirsen
  Interventions: Drug: Eteplirsen
- Golodirsen
  Interventions: Drug: Golodirsen
- Casimersen
  Interventions: Drug: Casimersen

INTERVENTIONS:
Drug: Eteplirsen — No study medication will be provided by the Sponsor as a condition to participate in this observational study, and all decisions concerning each participant's treatment are at the discretion of the participant's treating physician. Participants will receive treatment as prescribed by the treating physician as part of standard of care.
  Other Names: AVI-4658; EXONDYS 51; EXONDYS
  Groups: Eteplirsen
Drug: Golodirsen — No study medication will be provided by the Sponsor as a condition to participate in this observational study, and all decisions concerning each participant's treatment are at the discretion of the participant's treating physician. Participants will receive treatment as prescribed by the treating physician as part of standard of care.
  Other Names: SRP-4053; VYONDYS 53
  Groups: Golodirsen
Drug: Casimersen — No study medication will be provided by the Sponsor as a condition to participate in this observational study, and all decisions concerning each participant's treatment are at the discretion of the participant's treating physician. Participants will receive treatment as prescribed by the treating physician as part of standard of care.
  Other Names: SRP-4045; AMONDYS 45
  Groups: Casimersen

SUMMARY:
This is a phase 4, multicenter, prospective, observational study designed to collect both medical history data and prospective data on Duchenne Muscular Dystrophy (DMD) treatment outcomes in participants receiving eteplirsen, golodirsen, and casimersen in routine clinical practice. Participants in this study will have been prescribed eteplirsen, golodirsen, or casimersen commercially prior to entry into the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Is willing to provide informed assent or consent (if applicable) and has a parent(s) or legal guardian(s) or is a participant ≥18 years of age who is (are) willing to provide informed consent for the participant to participate in the study and comply with study data collection procedures.
* Has an established clinical diagnosis of DMD, as documented prior to screening by a genetic report.
* Receiving, or initiating treatment with, eteplirsen, golodirsen, or casimersen at the time of observational study enrollment. Note: Participants with a prescription for eteplirsen, golodirsen, or casimersen at enrollment must initiate the exon-skipping therapy within 6 months of the date of enrollment or will no longer be eligible for this study. Note: Enrollment of eteplirsen participants has been completed, no additional participants will be enrolled.

Key Exclusion Criteria:

* Is currently participating in any DMD interventional study at the time of this study enrollment.
* Has declined to provide consent for collection of their genetic data.
* Has a medical condition or confounding circumstances that, in the opinion of the Investigator, might compromise:

  1. The participant's ability to comply with the protocol-required procedures
  2. The participant's wellbeing or safety, and/or
  3. The clinical interpretability of the data collected from the participant.

Other inclusion/exclusion criteria may apply.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants within each prescriber's practice who are receiving eteplirsen, golodirsen, or casimersen, in routine clinical practice, and who meet the study eligibility criteria and provide informed consent (either by the participant or through authorization by a legal guardian), will be invited to enroll into the study and will be followed according to the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Loss of Ambulation (LOA) | Up to 5 years
Time to Rise From the Floor (Supine to Stand) | Up to 5 years
Time to Walk/Run 10 Meters | Up to 5 years
Performance of Upper Limb Module for DMD 2.0 (PUL 2.0) Entry Item A | Up to 5 years
Pulmonary Function, as Measured by Forced Vital Capacity (FVC) (% Predicted) | Up to 5 years
Cardiac Function, Including Left Ventricular Ejection Fraction (LVEF) as Measured by Echocardiogram (ECHO) | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center - PIN, New York, New York
  - Duke Lenox Baker Children's Hospital, Durham, North Carolina
  - Atrium Health Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Cook Children's Hospital, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - UVA Children's Hospital, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington